CLINICAL TRIAL: NCT07243002
Title: Real-world Evaluation of Patient Outcomes and Experiences With Ribociclib Early Adopters: A Hybrid Study With Prospective Patient-reported Outcomes and Retrospective Clinical Chart Review.
Brief Title: Real-world Evaluation of Patient Outcomes and Experiences With Ribociclib Early Adopters.
Acronym: REPOWER
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011O12005
Record Dates: First submitted 2025-11-13; First posted 2025-11-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: ribociclib, abemacicblib; Breast Cancer; Non interventional study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (2):
- Ribociclib arm: Patient treated with ribociclib and Endocrine Therapy (ET) per standard of care
- Abemaciclib arm: Patient treated with abemaciclib and Endocrine Therapy (ET) per standard of care

SUMMARY:
This non-interventional study (NIS) aims to evaluate effectiveness, persistence, treatment patterns, adverse events (AEs), and patient-reported experience (including adherence, treatment satisfaction, health-related quality of life [HRQoL], work productivity, and etc.), among HR+/HER2- stage II and III eBC patients treated with ribociclib + ET, and to evaluate AEs and patients-reported experience among HR+/HER2- stage II and III eBC patients treated with abemaciclib + ET, as per local label.

DETAILED DESCRIPTION:
This will be a multi-center, multi-country, observational, non-interventional, hybrid study among HR+/HER2- stage II or III eBC patients treated with ribociclib + ET or abemaciclib + ET, as per local label in routine clinical care settings.

The study will include a retrospective and a prospective part. The hybrid design will combine retrospective data extraction from patients' EHRs and prospective data collection from validated PRO questionnaires, bespoke questions, and qualitative interviews, to provide comprehensive data on the patient population.

The exploratory objectives will assess HR+/HER2- stage II and III eBC patients treated with abemaciclib + ET. No formal comparison between the cohorts will be made

ELIGIBILITY:
Inclusion Criteria:

* Males or females.
* Diagnosed with breast cancer, as defined by the International Classification of Diseases (ICD), 9th or 10th Revision, Clinical Modification (ICD-9-CM 174.xx, 175.xx/ICD-10-CMC50.xx).
* Aged ≥18 years (or local legal age of consent) at the date of initial breast cancer diagnosis.
* Patients with anatomic staging II and III as determined using American Joint Committee on Cancer (AJCC) Criteria.
* Have initiated adjuvant therapy with ribociclib or abemaciclib, per the approved local label, in combination with ET (within 14 days prior to enrollment).
* Have HR+ status, as determined by the closest biomarker test on or before the adjuvant therapy initiation date:

  * Tested positive for estrogen receptor (ER+), or
  * Tested positive for progesterone receptor (PR+), or
  * Tested positive for both.
* Tested negative for HER2 (HER2-) using the closest biomarker test on or before the adjuvant therapy initiation date.

Exclusion Criteria:

* Patients with local or distant breast cancer recurrence before the ribociclib/abemaciclib initiation date.
* Patients enrolled in clinical trials (receiving treatment with clinical study drugs in any setting, i.e., neoadjuvant, adjuvant, local/regional, metastatic) during the 12-month baseline period.
* Patients physically/mentally incapable of understanding the study requirements or fulfilling data collection instruments and require the support of a legally authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early breast cancer stage II or III, ER+ or PR+ (or both) and HER2-, treated per standard of care with ribociclib plus Endocrine Therapy (N=2650) or abemaciclib plus Endocrine Therapy (N=250).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2030-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (iDFS) | 36 months
  iDFS is defined as time to first invasive breast cancer recurrence (ipsilateral, contralateral, local/regional, distant), new primary invasive cancer, or death from breast cancer, non-breast cancer or unknown cause.
Distant disease-free survival (DDFS) | 36 months
  Distant disease-free survival (DDFS) is defined as time to first distant recurrence, second primary invasive cancer, or death from breast cancer, non-breast cancer or unknown cause.
  This will be assessed based on STEEP criteria version 2.0 (Standardized Definitions for Efficacy End Points in Adjuvant Breast Cancer Trials) and collected retrospectively from patient chart.

SECONDARY OUTCOMES:
Adherence to ribociclib + ET assessed using the MARS-5 tool | Up to approximately 36 months
  The MARS-5 (Medication Adherence Report Scale) is a 5 item questionnaire designed to assess patient adherence to treatment. Score is ranging from 1 (always) to 5 (never) for each item. The total score ranges from 5 to 25, where a higher MARS-5 score indicates higher adherence. One item assesses unintentional non-adherence, and four items assess intentional non-adherence.
Adherence to ribociclib + ET assessed using bespoke questions. | Up to approximately 36 months
  6 bespoke questions as to adherence have been added to capture key behavior patterns (ie, use of other products, cost, schedule, time, access to medication and convenience). Score is ranging from 1 (always) to 5 (never) for each item.
Treatment satisfaction with ribociclib + ET assessed using bespoke questions. | Up to approximately 36 months
  Treatment satisfaction will be assessed using 8 bespoke questions, focusing on key domains such as expectations, feelings about side effects, management of side effects, and overall satisfaction. Responses are scored on a 5-point Likert scale ranging 1 (always) to 5 (never) depending on satisfaction level.
Changes in Health Related Quality of Life (HRQoL) with ribociclib + ET assessed using EORTC QLQ-C30. | Up to approximately 36 months
  Health related quality of life will be assessed with the EORTC QLQ c30, which was designed to measure psychical, social, emotional, cognitive functions, symptom and health status in individuals with cancer.
  Item 1-28 are scored on a 4 point Liker t scale (1 + not at all, to 4 + very much). Item 29 and 30 are scored on a 7 point numerical rating scale (from 1 + very poor to 7 + Excellent).
  Raw scored are transformed and standardized with scores ranging from 0 to 100. A higher score represents either a better functioning, a higher level of Quality of life or a worse (higher) level of symptomatology.
Changes in Health Related Quality of Life (HRQoL) with ribociclib + ET assessed using EORTC QLQ-BR42. | Up to approximately 36 months
  The EORTC QLQ BR42 is a specific breast cancer questionnaire to be used in conjunction with the EORTC QLQ c30. Items were designed to measure treatment side effect, symptoms, body image sexual functioning, breast satisfaction, future perspective, sexual enjoyment and weight gain.
  All items are scored on a 4-point Likert scale (from 1 = Not at all, to 4 = Very much). Items and domains are transformed and scores range between 0-100. Higher scores represent higher (better) functioning or higher levels (worse) symptomatology .
Changes in Long Term Health Related Quality of Life (HRQoL) with ribociclib + ET assessed using bespoke questions. | Up to approximately 36 months
  Health related quality of life assessed using bespoke questions to evaluate long term quality of life.
  Three bespoke questions were designed to measure long term QoL. The questions will be scored individually from 1 (Always) to 5 (Never), scores will be reversed as needed.
  There are also 2 bespoke questions to assess the impact on cognitive functions, both are scored individually from 1 (Always) to 5 (Never) with higher score indicating better cognitive functions.
Work productivity measured using WPAI | Up to approximately 36 months
  This is assessed using the WPAI tool, focusing on key aspects such as absenteeism, presenteeism, work productivity loss, activity impairment, and long-term impact of side effects on work activity.
  This questionnaire has 6 questions, which are used to calculate 4 types of scores, which are absenteeism (work time missed), presenteeism (impairment at work/reduced on the job effectiveness), work productivity loss (overall work impairment), and activity impairment. The scores are expressed in percentage with higher numbers indicating greater impairment and less productivity.
Patients' experience of treatment in HR+/HER2- stage II and III eBC patients treated with ribociclib + ET | Up to approximately 12 months
  Patients' experience of treatment assessed using qualitative interviews conducted in the sub-cohort of ribociclib + ET in the US only.
Work productivity in HR+/HER2- stage II and III eBC patients treated with ribociclib + ET using bespoke questions. | Up to approximately 36 months
  One bespoke question is used to evaluate impact of side effect on work productivity. The question is rated from 1 (always) to 5 (never) with higher score indicating better situation (reduced impact on work).
Persistence to ribociclib + ET | Up to approximately 36 months
  Proportion of patients who continue (persist) and discontinue ribociclib + ET.
Distant disease-free survival | At 12, 24 and 36 months
  Distant disease-free survival (DDFS) is defined as the time to first distant recurrence, second primary invasive cancer, or death from breast cancer, non-breast cancer or unknown cause.
Overall survival | At 12, 24 and 36 months
  Overall survival (OS) is defined as time to death from breast cancer, non-breast cancer or unknown cause.
Distant recurrence-free survival | At 12, 24 and 36 months
  Distant recurrence-free survival (DRFS) is defined as the time to first distant recurrence or death from breast cancer, non-breast cancer or unknown cause.
Invasive disease-free survival | At 12, 24 and 36 months
  Invasive disease-free survival (iDFS) is defined as the time to first invasive breast cancer recurrence (ipsilateral, contralateral, local/regional, distant), new primary invasive cancer, or death from breast cancer, non-breast cancer or unknown cause.
Invasive breast cancer-free survival | At 12, 24 and 36 months
  Invasive breast cancer-free survival (iBCFS) is defined as time to first invasive breast cancer recurrence (ipsilateral, local/regional, contralateral or distant) or death from breast cancer, non-breast cancer or unknown cause.
Patient and tumor characteristics at/around recurrence for HR+/HER2- stage II and III eBC patients treated with ribociclib + ET. | From index date until death, lost to follow-up, end of study period, or enrollment in clinical trials, whichever occurs first. The maximum follow-up time is expected to be up to 54 months
  Patient characteristics and tumor characteristics at/around recurrence, as available from chart.
AEs affecting HR+/HER2- stage II and III eBC patients treated with ribociclib + ET | Every 6 months until death, lost to follow-up, end of study period, or enrollment in clinical trials, whichever occurs first. Up to approximately 54 months
  AEs will be collected retrospectively from chart with their grading.
Number of participants by treatment patterns assessed in both the adjuvant and metastatic settings | From index date until death, lost to follow-up, end of study period, or enrollment in clinical trials, whichever occurs first. The maximum follow-up time is expected to be up to 54 months
  * Adjuvant setting: neoadjuvant, adjuvant, and any chemotherapy, type of primary site surgery, neoadjuvant ET, neoadjuvant chemotherapy and/or ET, type of ET, and TTD from adjuvant ribociclib initiation.
  * Metastatic setting: number of patients who receive 1L, most common treatment regimens at 1L, and TTD from the start of 1L following the first metastatic recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No